CLINICAL TRIAL: NCT04433624
Title: Analgesic Efficacy of the Erector Spinae Plane Block Using Bupivacaine Versus Bupivacaine/Magnesium Sulphate in Patients Undergoing Lumbar Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, doaa rashwan, Assistant professor Doaa Rashwan, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMBSUREC/07062020/Abd El Badei
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (B) (Active Comparator): will receive The bilateral ESP blocks before surgery
  Interventions: Other: Group (B)
- Group B MG (Active Comparator): will receive bilateral ESP blocks performed by each side) before surgery
  Interventions: Other: Group (B)

INTERVENTIONS:
Other: Group (B) — Group (B) (n=15): will receive The bilateral ESP blocks were performed by injecting 40 mL of 0.25% bupivacaine (20 mL into each side) into the fascial plane between the deep surface of the erector spinae muscle and the transverse processes of the lumbar vertebrae

SUMMARY:
Introduction:

Severe postoperative pain following spine surgery is a significant cause of morbidity, extended length of facility stay, and marked opioid usage

The analgesic regime for postoperative pain usually includes paracetamol,NSAIDs and opioids. The opioid epidemic as well as the opioid side effects2 (sedation,respiratory depression, constipation, delayed patient mobilization) has led perioperative physicians to find a way of decreasing the use of opioids. Increasing the use of regional anesthesia is one of the measures to this end. Ultrasound-guided erector spinae plane block (ESP) is a-- popular, interfascial regional technique that was initially described for the management of thoracic neuropathic pain . As the erector spinae fascia extends from the nuchal fascia cranially to the sacrum caudally, local anesthetic agents extend through several levels, and the block can be effective over a large area The ESP block provides effective postoperative analgesic effect for 24 hours in patients undergoing lumbar spinal surgery Magnesium sulfate (MGS) is a noncompetitive antagonist of N-methyl, D-aspartate (NMDA) receptors with an analgesic effect and is essential for release of acetylcholine from the presynaptic terminals and, similar to calcium channel blockers (CCB), can prevent the entry of calcium into the cell It is suggested that magnesium has many important roles to play in nociception

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of the Erector Spinae Plane Block using bupivacaine versus bupivacaine/magnesium sulphate in Patients Undergoing Lumbar Spine surgery

Inclusion criteria:

orthopedic and neurological patients undergoing posterior lumbar spine fusion [American Society of Anesthesiologists (ASA) physical status 1 or 2.

Exclusion Criteria:

1. -Contraindications for regional blocks (eg. Patient refusal Infection at the injection site, coagulopathy)
2. allergic reaction to drugs.
3. Patients with a history of liver, renal, heart and vascular failure, cardiac conduction disturbance.
4. opium addiction, any drug or substance abuse and chronic treatment with opium, non-steroidal anti-inflammatory drugs and calcium channel blockers (CCB).

The patients will be blinded to the study drugs and will be randomly assigned into two equal groups by opaque sealed envelope as follows:

Group (B) (n=15): will receive The bilateral ESP blocks were performed by injecting 40 mL of 0.25% bupivacaine (20 mL into each side) into the fascial plane between the deep surface of the erector spinae muscle and the transverse processes of the lumbar vertebrae

Group B MG (n=15): will receive bilateral ESP blocks performed by each side) and and 500 mg magnesium sulphate into the fascial plane between the deep surface of the erector spinae muscle and the transverse processes of the lumbar vertebrae for pain management after lumbar spinal surgery injecting 40 mL of 0.25% bupivacaine(20 mL into each side)

ELIGIBILITY:
Inclusion Criteria:

* orthopedic
* neurological patients
* undergoing posterior lumbar spine fusion
* American Society of Anesthesiologists (ASA) physical status 1 or 2.

Exclusion Criteria:

* Contraindications for regional blocks
* allergic reaction to drugs.
* Patients with a history of liver, renal, heart and vascular failure, cardiac conduction disturbance.
* opium addiction, any drug or substance abuse and chronic treatment with opium, non-steroidal anti-inflammatory drugs and calcium channel blockers (CCB).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-18 (Estimated); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
time to first request of analgesics in hours | change from base line for 24 hours
  time to first request of analgesics by the pateint in hours

CONTACTS AND LOCATIONS:
Locations (1):
- Banī Suwayf, Egypt, 11391, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided